CLINICAL TRIAL: NCT06914947
Title: Brain Health Together: Use of Human-centered Design to Develop and Pilot a Virtual Group Brain Health Program
Brief Title: Brain Health Together: Development and Pilot Test
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: R44AG074727-B; R44AG074727 (NIH)
Record Dates: First submitted 2025-04-04; First posted 2025-04-07 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Impairment; Subjective Cognitive Decline; Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-arm Pilot: 12-week pilot study with data collection and analysis at the completion of the initial 4 weeks of the program and at the completion of 12 weeks.
  Interventions: Behavioral: Brain Health Together

INTERVENTIONS:
Behavioral: Brain Health Together — Each week, the program included a 1-hour group brain health education class, a 1-hour group Moving Together class, and a 30-minute individual brain health coaching session (total: 2.5 hours/week). Before the first session, participants were asked to complete a brief online survey about lifestyle behaviors and medical conditions related to dementia risk. The first 4 brain health education classes focused on general content to introduce and reinforce the concept that healthy lifestyle behaviors and management of chronic medical conditions can improve cognitive function, delay cognitive decline, and potentially prevent dementia. Another goal was to introduce participants to health coaching and to help participants each set specific, measurable, achievable, realistic, time-limited (SMART) goals to improve brain health. The remaining 8 weeks were adjusted to accommodate participant feedback in the early portion of the pilot study.

SUMMARY:
The objectives of this study were to develop and pilot-test Brain Health Together (BHT), a 12-week, virtual-group program that combines our evidence-based, mind-body, group movement program with brain health education and coaching to reduce dementia risk through targeting modifiable risk factors among older adults with cognitive impairment.

DETAILED DESCRIPTION:
Our study design for developing, pilot-testing, and refining the BHT program was conducted in 2 phases. In Phase 1, the investigators used a human-centered design approach to deeply understand and respond to the needs, challenges, and motivations of potential users when developing the BHT program. In Phase 2, the investigators performed a pilot study to refine BHT program content and assess acceptability and potential feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment or subjective cognitive decline
* English language proficiency
* Active participants in Moving Together (Intervention Arm)

Exclusion Criteria:

* wheelchair user
* medical condition, physical limitation, visual or hearing impairment or psychiatric condition that could affect ability to participate in a virtually-delivered multicomponent intervention
* moderate/severe dementia severity

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Our study population included people who were active participants in the Moving Together program as well as a purposeful sample of individuals who were not familiar with the Moving Together program. Together these individuals' perceptions would facilitate further examination and identification of challenges in understanding and managing MCI.
  Pilot Inclusion Criteria:
  * Mild cognitive impairment or subjective cognitive decline
  * English language proficiency
  * Active participants in Moving Together (Intervention Arm)
  Pilot Exclusion Criteria:
  * wheelchair user; medical condition, physical limitation, visual or hearing impairment or psychiatric condition that could affect ability to participate in a virtually delivered multicomponent intervention
  * moderate/severe dementia severity
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility | 12 weeks
  To examine feasibility, the investigators tracked participant attendance, calculated as the mean±standard deviation (SD) of sessions completed by each participant.
Acceptability | 12 weeks
  The investigators asked participants how likely they are to recommend BHT to others on a scale from 0 (not at all likely) to 10 (extremely likely) and calculated a net promoter score as the percentage of promoters (scores of 9 or 10) minus the percentage of detractors (scores of 0 to 6).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Given the small number of participants and the exploratory nature of this trial, participants could potentially be identifiable.